CLINICAL TRIAL: NCT06203912
Title: A Phase Ib Study of TGFbi NK Cells and Isatuximab for Myeloma Relapsed/Refractory to BCMA Targeting Therapy
Brief Title: Donor Immune Cells (TGFbi NK Cells) and Isatuximab for the Treatment of Relapsed or Refractory Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Elvira Umyarova (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor-Investigator, Elvira Umyarova, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-23093; NCI-2023-09969 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-12-12; First posted 2024-01-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Specimen Handling; Biopsy; Cyclophosphamide; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; isatuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cyclophosphamide, dexamethasone, TiNK, isatuximab) (Experimental): Patients receive cyclophosphamide IV on day 1, dexamethasone PO on days 1-4, TiNK IV on day 8, and isatuximab IV on days 8 and 15 of each cycle. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo bone marrow aspiration and biopsy during screening and on study, as well as optionally during follow up. Patients undergo ECHO during screening and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Drug: Cyclophosphamide; Drug: Dexamethasone; Procedure: Echocardiography; Biological: Isatuximab; Other: Questionnaire Administration; Biological: Universal Donor Expanded TGF-beta-imprinted NK Cells

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow aspiration and biopsy
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B-518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719; WR-138719
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Procedure: Echocardiography — Undergo echocardiography
  Other Names: EC
Biological: Isatuximab — Given IV
  Other Names: Hu 38SB19; Isatuximab-irfc; SAR 650984; SAR-650984; SAR650984; Sarclisa
Other: Questionnaire Administration — Ancillary study
Biological: Universal Donor Expanded TGF-beta-imprinted NK Cells — Given IV
  Other Names: Allogeneic TGFBi Expanded NK Cells; UD TGF-betai NK Cells; Universal Donor TGF-beta Imprinted Expanded NK Cells

SUMMARY:
This phase I trial tests the side effects and best dose of TGFbi natural killer (NK) cells (TiNK) when given together with isatuximab for the treatment of patients with multiple myeloma that has come back after a period of improvement (relapsed) or that has not responded to treatment (refractory). NK cells are a type of white blood cell that are known to spontaneously attack cancer cells. TiNK are NK cells made in a laboratory to have a higher response to tumor cells. A monoclonal antibody is a type of protein that can bind to certain targets in the body, such as molecules that cause the body to make an immune response (antigens). Immunotherapy with monoclonal antibodies, such as isatuximab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Patients also receive standard treatment (cyclophosphamide and dexamethasone) on this trial. Cyclophosphamide is in a class of medications called alkylating agents. It works by damaging the cell's DNA and may kill cancer cells. It may also lower the body's immune response. Dexamethasone is in a class of medications called corticosteroids. It is used to reduce inflammation and lower the body's immune response to help lessen the side effects of chemotherapy drugs. Giving TiNK and isatuximab with standard treatment may be a safe and effective treatment for relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and tolerability of transforming growth factor beta imprinted natural killer cells (TiNK) and isatuximab in patients with multiple myeloma (MM) relapsed or refractory (R/R) to BCMA-targeting therapy.

SECONDARY OBJECTIVES:

I. To evaluate the objective response rate (ORR) by International Myeloma Working Group (IMWG) criteria of TiNK and isatuximab in patients with MM R/R to BCMA-targeting therapy.

II. To determine the time to response (TTR), time to next therapy (TTNT), the duration of response (DOR), progression free survival (PFS), and overall survival (OS) at 1 year.

III. To determine correlatives of outcomes. IV. To assess quality of life (QOL) with therapy.

OUTLINE: This is a dose-escalation study of TiNK followed by a dose-expansion study.

Patients receive cyclophosphamide intravenously (IV) on day 1, dexamethasone orally (PO) on days 1-4, TiNK IV on day 8, and isatuximab IV on days 8 and 15 of each cycle. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo bone marrow aspiration and biopsy during screening and on study, as well as optionally during follow up. Patients undergo echocardiography (ECHO) during screening and blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 30 days, 60 days. Patients who discontinue study treatment for reasons other than progressive disease follow up every 12 weeks for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older with evidence of relapsed or refractory disease as defined by IMWG criteria and measurable disease as defined by any of the following:

  * Serum M-protein ≥ 0.5 g/dl
  * Urine monoclonal protein ≥ 200 mg/24h
  * Involved free light chain (FLC) level ≥ 10mg/dl (≥ 100mg/l) and an abnormal serum free light chain ratio (< 0.26, or > 1.65)
* Patients must have had at least 3 prior lines of therapy including lenalidomide, proteasome inhibitor (PI), anti-CD38 or anti-SLAMF7 directed antibody, and BCMA-targeting therapy.

  * Prior daratumumab or isatuximab is permitted but not in the immediate line prior to study entry
  * Prior autologous hematopoietic cell transplant is permitted
  * Prior allogeneic transplant is excluded
* Refractory (progressed on or within 60 days of treatment) to their last treatment

  * If chimeric antigen receptor t cell (CAR-T) therapy was the immediately prior therapy, then the definition of refractory disease will not be limited to within 60 days
  * Patients must be off last treatment for at least 2 weeks by the beginning of treatment on this protocol
* Hemoglobin ≥ 7g/dL
* Absolute neutrophil count (ANC) ≥ 1000/µL
* Platelets ≥ 70,000/µL

  * If plasma cell percentage on bone marrow biopsy core is > 30%, platelet requirement will be adjusted to 50,000/µl
* Total bilirubin < 2 mg/dL
* Aspartate aminotransferase (AST)/ alanine aminotransferase (ALT)/ alkaline phosphatase < 2.5 X the upper limit of normal (ULN)
* Calculated creatinine clearance of ≥ 30ml/min using Modification of Diet in Renal Disease (MDRD) formula
* Left ventricular ejection fraction ≥ 30%; baseline echocardiography (ECHO) is not required if ECHO was done within the preceding one year and patients do not have new signs/symptoms suggestive of heart failure
* No uncontrolled arrhythmias
* No New York Heart Association class III-IV heart failure
* 12-lead electrocardiogram (ECG) with QT interval calculated by Fridericia Formula (QTcF) interval of ≤ 470 msec
* Patients must provide informed consent
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of ≤ 2
* Fertility requirements:

  * Women of child bearing potential (WOCBP) must commit to either abstain continuously from heterosexual sexual intercourse or to use 2 methods of reliable birth control simultaneously. This includes one highly effective form of contraception (tubal ligation, intrauterine device [IUD], hormonal [birth control pills, injections, hormonal patches, vaginal rings or implants] or partner's vasectomy) and one additional effective contraceptive method (male latex or synthetic condom, diaphragm, or cervical cap). Contraception must begin 4 weeks prior to dosing and continue to 6 months after study treatment ending. Reliable contraception is indicated even where there has been a history of infertility, unless due to hysterectomy.
  * Investigators shall counsel WOCBP and male participants who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy
  * A negative pregnancy test will be required for all WOCBP within 24 hours before starting treatment drugs
  * Breast feeding is not permitted
  * Male patients must agree to use an adequate method of contraception (latex or synthetic condom) for the duration of the study and up to 6 months after study treatment ending
  * Criteria also applies to azoospermic males
  * Males should refrain from sperm donation during this time and continue for 6 months after study treatment ending

Exclusion Criteria:

* Patients with active (untreated or relapsed) central nervous system (CNS) MM
* Patients with Waldenstrom macroglobulinemia, primary AL amyloidosis, primary plasma cell leukemia, or polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes (POEMS) syndrome

  * Patients with secondary plasma cell leukemia are permitted
* Patients receiving concurrent corticosteroids at the time protocol therapy is initiated other than for physiologic maintenance treatment
* Concurrent use of complementary or alternative medicines that would confound the interpretation of toxicities and antitumor activity of the study drugs
* Patients with contraindications or allergy to cyclophosphamide and/or daratumumab/isatuximab
* Unacceptable respiratory risk factors defined by any one of the following criteria:

  * Chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) less than 50% of predicted normal
  * Moderate or severe persistent asthma within the past 2 years, or currently has uncontrolled asthma of any classification
* Unacceptable cardiac risk factors defined by any of the following criteria:

  * Complete left bundle branch, bifascicular block or clinically significant abnormal electrocardiogram (EKG) finding at screening
  * Congenital long QT Syndrome
  * Myocardial infarction or unstable angina within 6 months
* Patients who have received targeted or investigational agents within 2 weeks or within 5 half-lives of the agent and active metabolites (whichever is shorter) and who have not recovered from side effects of those therapies
* Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from the side-effects of surgery
* Patients with known positivity for human immunodeficiency virus (HIV) or active hepatitis B/C

  * Patients with chronic hepatitis B infection may be enrolled but must be provided prophylaxis (ex. entecavir for one year from start of therapy)
* Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention, other than non-melanoma skin cancer and carcinoma in situ of the cervix or breast, should not be enrolled
* Patients with any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to them by the study staff
* Any other medical condition, including mental illness or substance abuse, deemed by the investigator(s) to likely interfere with the patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results
* Life expectancy of 6 months or less

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AE) | Up to 60 days after completion of study treatment
  Will use the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 for AE collection. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns. The incidence of severe (grade 3+) adverse events or toxicities will be described. We will also assess tolerability of the regimen through assessing the number of patients who required dose modifications and/or dose delays. In addition, we will capture the proportion of patients who go off treatment due to adverse reactions.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years after completion of study treatment
  Will be defined as the total number of subjects whose best response is partial response (PR) or better divided by the number of patients. Will be reported overall with 95% binomial exact confidence intervals. Comparison of ORR among patient subgroups will be conducted using Fisher exact test.
Time to response | From start of treatment until measurement criteria are first met for PR, very good partial response (VGPR), or complete response (CR), assessed up to 2 years after completion of study treatment
  Cumulative incidence rates will be calculated and compared using Gray's test accounting for competing risks.
Time to next therapy | From start of treatment until initiation of the next line of therapy, assessed up to 2 years after completion of study treatment
  Cumulative incidence rates will be calculated and compared using Gray's test accounting for competing risks.
Duration of response | From the time measurement criteria are first met for PR or better (whichever status is recorded first) until the first date of progressive disease or death, assessed up to 2 years after completion of study
  Will be computed for subjects whose best response is either PR, VGPR, or CR. Will be analyzed using the Kaplan-Meier method.
Progression free survival | From start of treatment until disease progression or death, at 1 year
  Will be analyzed using the Kaplan-Meier method.
Overall survival | From start of treatment to the date of his or her death, at 1 year
  Will be analyzed using the Kaplan-Meier method.
Change in quality of life (QOL) using PROMIS G10 | Baseline up to 60 days after completion of study treatment
  Using the Patient-Reported Outcomes Measurement Information System Global 10 Quality of Life Survey (PROMIS G10 QOL) A repeated measures linear mixed model will be fit to all QOL scores. The response options are presented as 5-point (and single 11-point for pain rating scales). The results of the questions are used to calculate two summary scores.
Change in quality of life (QOL) using EORTC QLQ-MY20 | Baseline up to 60 days after completion of study treatment
  Using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Multiple Myeloma20 (EORTC QLQ - MY20). A repeated measures linear mixed model will be fit to all QOL scores. This incorporates four multi-item scales to assess disease symptoms, side effects of treatment, future perspective and body image. All of the scales and single-item measures range in score from 0 to 100. A high score for the symptom scales represents a high level of symptomatology or problems, whereas a high score for the functional scale represents a high level of functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Elvira Umyarova, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu